CLINICAL TRIAL: NCT02660515
Title: Operative Treatment of Intra-Articular Distal Radius Fractures With Versus Without Wrist Arthroscopy, a Randomized Controlled Trial
Brief Title: Operative Treatment of Intra-Articular Distal Radius Fractures With Versus Without Wrist Arthroscopy
Acronym: RADAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Collaborators: Erasmus Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Niels Schep, MD, PhD, Maasstad Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL54377.101.15
Record Dates: First submitted 2016-01-13; First posted 2016-01-21 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Distal Radius Fracture
Keywords: complete articular distal radius fracture; wrist arthroscopy
MeSH Terms: conditions — Wrist Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORIF (Active Comparator): The operation has to be performed within 3 weeks after the initial trauma. According to the current standard, antibiotic prophylaxis (Cefazoline, 1000 milligram intravenous) will be administered thirty minutes preoperatively. The distal radius will be approached according to Henry, which beholds an incision between the tendon of the flexor carpi radialis and the arteria radialis. After the fracture site is exposed, the fracture will be reduced and an appropriate volar locking plate will be positioned. The type and brand of the plate are at discretion of the treating surgeon. When a dorsal approach is deemed necessary the distal radius will be approached between the third and fourth dorsal extensor tendon compartments. To evaluate the quality of articular reduction, fluoroscopic images will be obtained. Wound closure will be performed using standard techniques.
  Interventions: Procedure: ORIF
- ORIF with additional wrist arthroscopy (Active Comparator): Surgery will be performed by a certified trauma surgeon, with experience in wrist arthroscopy. A delay of minimal 5 days before performing arthroscopy is mandatory to enable visualisation due to the organisation of the hematoma. During wrist arthroscopy, the forearm will be positioned upright and in neutral position, the elbow flexed by 90° and axial traction of 4-6 kg will be performed. Four portal entrees are created by superficial stab incisions and blunt preparation through the joint capsule; one midcarpal radiair and one midcarpal ulnar portal and the 3-4 and 6-R portal. A shaver is used for removal of fracture haematoma and osteocartilaginous debris. Cartilage damage will be graded using the Outerbridge classification system. With the 1 mm hook probe assessment of the quality of reduction and ligamentous injuries (TFCC, scapholunate and lunotriquetral) will be performed. Wound closure will be performed using standard techniques.
  Interventions: Procedure: Additional wrist arthroscopy; Procedure: ORIF

INTERVENTIONS:
Procedure: Additional wrist arthroscopy
  Arms: ORIF with additional wrist arthroscopy
Procedure: ORIF
  Other Names: open reduction and internal fixation

SUMMARY:
Open reduction and internal fixation of intra-articular distal radius fractures leads to better functional outcomes the first 6 months compared to non-operative treatment. However, some patients continue to have a painful and stiff wrist post-operatively. Arthroscopically assisted removal of intra- articular fracture haematoma and debris may reduce pain and improve the functional outcomes following operative treatment of intra-articular distal radius fractures. Moreover, during arthroscopy the quality of the reduction and the presence of associated ligamentous injuries can be assessed. Therefore the objective of this study is to compare the functional outcome of internal plate fixation with additional wrist arthroscopy versus conventional fluoroscopic assisted internal plate fixation in adult patients with displaced intra-articular distal radius fractures.

DETAILED DESCRIPTION:
Distal radius fractures account for 17% of all fractures seen at the emergency department. Fifty percent of these fractures are intra-articular. The past several years an increase in open reposition internal fixation (ORIF) for distal radius fractures has been observed. This technique leads to a quicker resume of function the first 3 to 6 months compared to non-operative treatment. However, some patients continue to have a painful and stiff wrist postoperatively. Arthroscopically assisted removal of intra-articular fracture haematoma and debris may improve the functional outcomes following operative treatment of intra-articular distal radius fractures. Moreover, during arthroscopy the quality of the reduction and the presence of associated ligamentous injuries can be assessed.

To our knowledge, no studies have been carried out to further examine the use of arthroscopy after internal plate fixation to remove fracture haematoma and debris on functional outcomes. Therefore, the purpose of this randomised controlled trial is to determine the difference in functional outcome, assessed with the Patient-Rated Wrist Evaluation (PRWE) score, after internal plate fixation with an additional wrist arthroscopy and conventional fluoroscopically assisted internal plate fixation in adult patients with displaced complete articular distal radius fractures. Secondary, we aim to determine the difference in functional outcomes with the Disability of the Arm, Shoulder and Hand (DASH) score, post-operative pain, range of motion, grip strength, complications, quality of life (SF-36), and cost-effectiveness. Additionally, for patients undergoing additional wrist arthroscopy the quality of reduction, associated ligamentous injuries and cartilage damage will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Displaced intra-articular distal radius fracture (AO/OTA type C) as classified on lateral, posterior anterior and lateral carporadial radiographs by a radiologist or trauma surgeon
* Inacceptable closed reduction requiring open reduction and internal fixation

Exclusion Criteria:

* Dorsal plate fixation in case the radiocarpal joint needs to be opened
* Patients with impaired wrist function prior to injury due to arthrosis/neurological disorders of the upper limb
* Open distal radius fractures
* Multiple trauma patients (Injury Severity Score (ISS) ≥16)
* Other fractures of the affected extremity (except from ulnar styloid process)
* Fracture of other wrist
* Insufficient comprehension of the Dutch language to understand a rehabilitation program and other treatment information as judged by the attending physician
* Patient suffering from disorders of bone metabolism other than osteoporosis (i.e. Paget's disease, renal osteodystrophy, osteomalacia)
* Patients suffering from connective tissue disease or (joint) hyperflexibility disorders such as Marfan's, Ehler Danlos or other related disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation | 3 months
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of three subscales: Pain, Function and Cosmetics.

SECONDARY OUTCOMES:
Disability of the Arm, Shoulder and Hand Disability of the Arm, Shoulder and Hand | 3 and 6 weeks, and 3, 6 and 12 months
  The Disabilities of the Arm, Shoulder and Hand (DASH) score is a 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb.
Pain | 1 day post-operative and 1, 3 and 6 weeks and 3 months
  Pain as indicated on a visual Analogue Scale (VAS), in which 0 implies no pain and 10 the worst possible pain. Patients will be asked to give an estimation of the type and quantity of pain medication taken during all follow-up visits.
Range of motion | 3 and 6 weeks and 3 months
  Range of motion of the wrist measured on both sides with a handheld goniometer.
Grip strength | 3 and 6 weeks and 3 months
  Grip strength as measured with a dynamometer.
Complications | 1 day post-operative and 1, 3 and 6 weeks and 3 months
  Complication rate such as: wound and/or plate infection, tendon irritation and/or rupture, neuropathy and the occurrence of complex regional pain syndrome.
Cost-effectiveness | 3 and 6 weeks and 3 months
  Cost-effectiveness and cost-utility measured with an economic evaluation questionnaire based on the EQ-6D and the Standard Form Health and Labour questionnaire.
  Cost-effectiveness and cost-utility measured with an economic evaluation questionnaire based on the EQ-6D and the Standard Form Health and Labour questionnaire.
Associated injuries | Peroperative
  In the intervention group the quality of reduction, associated ligamentous injuries and cartilage damage will be assessed. Ligamentous injuries are divided in TFCC injuries, classified according to the Palmer classification and scapholunate ligament and lunotruquetral injuries, graded according to the Geissler classification.
Patient Rated Wrist Evaluation | 3 and 6 weeks, and 6 and 12 months
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of three subscales: Pain, Function and Cosmetics.

CONTACTS AND LOCATIONS:
Locations (1):
- Maasstad Hospital, Rotterdam, Nederland, Netherlands

REFERENCES:
- [Derived] Mulders MAM, Selles CA, Colaris JW, Peters RW, van Heijl M, Cleffken BI, Schep NWL. Operative Treatment of Intra-Articular Distal Radius Fractures With versus Without Arthroscopy: study protocol for a randomised controlled trial. Trials. 2018 Feb 2;19(1):84. doi: 10.1186/s13063-017-2409-2. PMID 29394904